CLINICAL TRIAL: NCT01512927
Title: Electronic Stethoscope and Computer-aided Diagnostic System in Detecting Arteriovenous Fistula (AVF) Stenosis
Brief Title: Electro Stethoscope in Detect Arteriovenous Fistula (AVF) Stenosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 201112015RIC
Record Dates: First submitted 2012-01-15; First posted 2012-01-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Arteriovenous Fistula
Keywords: electronic stethoscope; arteriovenous fistula; hemodialysis,
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ESRD with regular hemodialysis

SUMMARY:
The incidence and prevalence of end-stage renal disease (ESRD) in Taiwan are both the highest worldwide from 2001 to 2008. In Taiwan, more than 90% of the ESRD patients are hemodialysis patients. Either arteriovenous fistula (AVF) or arteriovenous graft (AV graft) is essential for the vascular access of these patients. However, frequent AVF stenosis or thrombosis occurs in 10-30% hemodialytic patients, and the rates are even higher, around 30-70%, in those who has a past history of AVF/AV graft stenosis. Therefore, early detection of AVF stenosis is essential in caring for these hemodialysis patients in terms of medical economics and psychological impact. Unfortunately, angiographic study is expensive and invasive and needs contrast medium injection. The diagnostic accuracy of color duplex ultrasound in AVF stenosis remains satisfactory, but it is not always available when decreased AVF flow or an acute thrombotic event occurs. Continuous AVF/ AV graft flow monitoring by patient himself is a better option in terms of long-term care. Previous study indicated that stethoscope waveform analysis could be used as an alternative to diagnosis of vascular stenosis. Therefore, we aim to investigate AVF/ AV graft stenosis by using the electronic stethoscope (3M Littmann) for AVF sound recording, followed by software analysis by using waveform decomposition, principle component analysis (PCA) and sequential forward selection algorithm [xx]. Our study results will provide a new diagnostic option, which is low cost, non-invasive and self-monitoring, of AVF stenosis in ESRD patients.

DETAILED DESCRIPTION:
Hemodialysis is a well-established method for removal of fluid and uremic toxins and prolonging survival in patients with end-stage renal disease (ESRD). The most common permanent vascular assesses are autogenous and non-autogenous arteriovenous (AV) fistula, referred as AV fistula and AV graft, respectively. In Taiwan, both incidence and prevalence of ESRD remain highest worldwide. However, frequent vascular stenosis/ thrombosis events occurred because of repeated needle punctures. These will exert a large economic burden to our society and psychological impacts on ESRD patients [1]. Therefore, it is essential to develop an easy and patient-centered method to monitor the flow status in either AV fistula or AV graft.

Physical examination and auscultation are simple monitoring methods to assess the vascular access. There were several signs reported to be associated vascular stenosis, such as prolonged bleeding, arm edema, and changes in pulse characteristics of the vascular access, but they need a high level of skill and experience from the operator, such as doctors and nurses [2].

Unfortunately, angiographic study is expensive and invasive and needs contrast medium injection. The diagnostic accuracy of color duplex ultrasound in AVF stenosis remains satisfactory, but it is not always available when decreased AVF flow or an acute thrombotic event occurs. Continuous AVF/ AV graft flow monitoring by patient himself is a better option in terms of long-term care. Previous study indicated that stethoscope waveform analysis could be used as an alternative to diagnosis of vascular stenosis. Previous acoustic studies indicated that increased sound intensity, extra sounds, and higher spectral energy infrequency domain, ranging between 300 Hz and 1000 Hz. These findings are associated with the change from laminar flow to turbulent flow downstream the site of vascular stenosis [3]. In addition, phonoangiography studies pointed out that the systolic peak of stenotic segment is higher and narrower in the time domain compared to non-stenotic segment Methods: This is an observational cohort study. We plan to recruit 150 eligible patients with ESRD under regular hemodialysis for at least one year in national Taiwan University Hospital.

1. Data gathering A. The first group of patients (study group) will be recruited from hose referred to endovascular intervention, e.g. angioplasty, due to vascular access dysfunction (n=30). An electronic stethoscope (3M-Littmann) will be used to record digital sound signals at 5 points with 30 seconds each, including AV junction, proximal and distal to both needle puncture sites, respectively. All data will be transferred to a computer for further anlaysis.

   B. The second group (validation cohort) will be recruited from patients with regular hemodialysis (HD) and received angioplasty at National Taiwan University Hospital (n=120). Those patients who received angioplasty for AVF or AV graft stenosis will also received follow-up angiography 12 weeks after angioplasty. We will record digital AVF/AV graft sound signals as mentioned above. In addition, blood pressure and AVF/AVG venous pressure, heart rate will be recorded. Diameter stenosis of restenotic segment will also be recorded and a diameter stenosis of 50% is regarded as significant.
2. Post-processing The proposed method is based on the analysis of the envelope of the sound signals. Before, calculating the envelope, all signals will be down-sampled to 2k Hz, followed by a linear-phase, finite impulse response low-pass filter. PCA will then be applied to analysis as described previously [1-4]. PCA (principal components analysis)
3. Analysis Sensitivity, specificity and diagnostic accuracy will be calculated based on each diagnostic criteria or basal function. Area under ROC curve will be calculated based on each diagnostic criteria derived from PCA method.

ELIGIBILITY:
Inclusion Criteria:

1. Age is more than 20 year-old.
2. End-stage renal disease with regular hemodialysis for more than one year

Exclusion Criteria:

1. AVF/ AV graft is not located in upper arm.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Feng Yeih, Ph.D., Principal Investigator — No.7, Chung Shan S. Rd., Zhongzheng Dist., Taipei City 100, Taiwan (R.O.C.)
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan